CLINICAL TRIAL: NCT05072405
Title: Interactions of Herbs With Statin Drugs and Potential Mediation by Drug Transporters
Brief Title: The Interaction of Herbs and Statins
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Brian Tomlinson, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: herbals
Record Dates: First submitted 2021-08-29; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Drug Interaction
Keywords: Statins
MeSH Terms: interventions — Simvastatin; Tea; Soybean Proteins; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Open-label, single-dose, randomized, three-phase (no herbs, with green tea, with soy isoflavones), once with rosuvastatin and once with simvastatin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- simvastatin 20 mg (Zocor®, MSD) (Other): simvastatin 20 mg are given on 3 occasions: 1. without herbs; 2. with green tea extract containing EGCG 800 mg once daily for 14 days before statin dosing; 3. with soy isoflavones extract containing isoflavones 120 mg once daily for 14 days before statin dosing, with at least 4-week washout period between phases.
  Interventions: Drug: Simvastatin 20 mg (Zocor®, MSD)
- rosuvastatin 10 mg (Crestor®, Astra Zeneca) (Other): rosuvastatin 10 mg are given on 3 occasions: 1. without herbs; 2. with green tea extract containing EGCG 800 mg once daily for 14 days before statin dosing; 3. with soy isoflavones extract containing isoflavones 120 mg once daily for 14 days before statin dosing, with at least 4-week washout period between phases
  Interventions: Drug: rosuvastatin 10 mg (Crestor®, Astra Zeneca)

INTERVENTIONS:
Drug: Simvastatin 20 mg (Zocor®, MSD) — Simvastatin 20 mg given once alone, once with green tea extract and once with soy isoflavones extract.
  Other Names: Green tea extract; Soy isoflavones extract
  Arms: simvastatin 20 mg (Zocor®, MSD)
Drug: rosuvastatin 10 mg (Crestor®, Astra Zeneca) — rosuvastatin 10 mg are given once alone, once with green tea extract and once with soy isoflavones extract.
  Other Names: Green tea extract; Soy isoflavones extract
  Arms: rosuvastatin 10 mg (Crestor®, Astra Zeneca)

SUMMARY:
This project includes two separate pharmacokinetic studies with simvastatin and rosuvastatin, respectively. Each study is an open-label, single-dose, randomized, three-phase (no herbs, with green tea, with soy isoflavones) clinical pharmacokinetic study design with a wash-out of at least 4-weeks between phases. The aim is to examine whether green tea extract and soy isoflavones affect the pharmacokinetics of simvastatin and rosuvastatin in healthy subjects and whether these interactions are influenced by polymorphisms in the relevant drug transporters, solute carrier 1B1 (SLCO1B1) and adenosine triphosphate (ATP) binding cassette G2 (ABCG2) and to identify whether polymorphisms in drug transporters influence the pharmacokinetics of simvastatin and rosuvastatin. After informed consent is obtained, subjects are required to abstain from any prescription or non-prescription medications 2 weeks before and throughout the study. Subjects are given a single dose of simvastatin 20 mg (Zocor®, MSD) or rosuvastatin 10 mg (Crestor®, Astra Zeneca) on 3 occasions: 1. without herbs; 2. with green tea extract; 3. with soy isoflavones extract. The green tea extract and soy isoflavones extract are given at a dose containing epigallocatechin gallate (EGCG) 800 mg once daily or isoflavones 120 mg once daily for 14 days before statin dosing with at least 4-week washout period between phases. Blood samples are taken at intervals from 0 to 24 hours on the statin dosing days. During the study, subjects are reminded frequently of the requirements on diet.

DETAILED DESCRIPTION:
Healthy Chinese male subjects aged 18-45 years are recruited from a pool of over 200 healthy volunteers who had been genotyped for the SLCO1B1 388A>G, 521T>C and ABCG2 421C>A polymorphisms. All subjects are required to abstain from any prescription or non-prescription medications 2 weeks before and throughout the study. They are not allowed to take alcohol, tea, grapefruit juice, caffeine, soybean milk or dietary supplements and herbal products 2 weeks before and throughout the entire study period. They are also not allowed to smoke 2 weeks before and throughout the study. Subjects are requested to fast for 10 h before and 4 h after drug administration during the blood sampling sessions. Meals are standardized and consumed at 4 h and 10 h post dosing. Drinking water are not allowed from 1 h pre-dose to 1 h post-dose except that needed for drug dosing at the time of blood sampling sessions. Subjects are given a single dose of simvastatin 20 mg (Zocor®, MSD) or rosuvastatin 10 mg (Crestor®, Astra Zeneca) on 3 occasions: 1. without herbs; 2. with green tea extract; 3. with soy isoflavones extract. The green tea extract and soy isoflavones extract are given at a dose containing EGCG 800 mg once daily or isoflavones 120 mg once daily for 14 days before statin dosing with at least 4-week washout period between phases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese male subjects aged 18 - 45 years
* healthy volunteers who had been genotyped for the SLCO1B1 388A>G, 521T>C and ABCG2 421C>A polymorphisms.

Exclusion Criteria:

* Female
* Patients with any disease
* Volunteers who cannot follow the instructions
* Volunteers who don't sign the informed consent.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-01-11 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2021-08-28 (Actual)

PRIMARY OUTCOMES:
The interactions of green tea extract and soy isoflavones on the maximum plasma concentration of simvastatin | 14 weeks
  Maximum plasma concentration for simvastatin comparing: 1. without herbs; 2. with green tea extract; 3. with soy isoflavones extract.
The interactions of green tea extract and soy isoflavones on the area under plasma concentration-time curve of simvastatin | 14 weeks
  Area under plasma concentration-time curve for simvastatin comparing: 1. without herbs; 2. with green tea extract; 3. with soy isoflavones extract.
The interactions of green tea extract and soy isoflavones on the maximum plasma concentration of rosuvastatin | 14 weeks
  Maximum plasma concentration for rosuvastatin comparing: 1. without herbs; 2. with green tea extract; 3. with soy isoflavones extract.
The interactions of green tea extract and soy isoflavones on the area under plasma concentration-time curve of rosuvastatin | 14 weeks
  Area under plasma concentration-time curve for rosuvastatin comparing: 1. without herbs; 2. with green tea extract; 3. with soy isoflavones extract.

SECONDARY OUTCOMES:
The influence of polymorphisms in drug transporters on the maximum plasma concentration of simvastatin and the interaction with herbs. | 14 weeks
  Maximum plasma concentration for simvastatin comparing: 1. without herbs; 2. with green tea extract; 3. with soy isoflavones extract with subjects divided according to genotypes of drug transporters.
The influence of polymorphisms in drug transporters on the area under plasma concentration-time curve of simvastatin and the interaction with herbs. | 14 weeks
  Area under plasma concentration-time curve for simvastatin comparing: 1. without herbs; 2. with green tea extract; 3. with soy isoflavones extract with subjects divided according to genotypes of drug transporters.
The influence of polymorphisms in drug transporters on the maximum plasma concentration of rosuvastatin and the interaction with herbs. | 14 weeks
  Maximum plasma concentration for rosuvastatin comparing: 1. without herbs; 2. with green tea extract; 3. with soy isoflavones extract with subjects divided according to genotypes of drug transporters.
The influence of polymorphisms in drug transporters on the area under plasma concentration-time curve of rosuvastatin and the interaction with herbs. | 14 weeks
  Area under plasma concentration-time curve for rosuvastatin comparing: 1. without herbs; 2. with green tea extract; 3. with soy isoflavones extract with subjects divided according to genotypes of drug transporters.

CONTACTS AND LOCATIONS:
Overall Officials: BRIAN TOMLINSON, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong